CLINICAL TRIAL: NCT05338905
Title: Intensive Symptom Surveillance Guided by Machine Learning-Directed Risk Stratification (INSIGHT)
Brief Title: Intensive Symptom Surveillance Guided by Machine Learning-Directed Risk Stratification in Patients With Non-Metastatic Head and Neck Cancer, The INSIGHT Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: I 2272021; NCI-2022-01920 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 2272021 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2022-03-29; First posted 2022-04-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (quality of life questionnaire) (Experimental): Patients complete a quality of life questionnaires over 10-15 minutes BIW during standard of care radiation therapy and QW for the first month after completing standard of care radiation therapy course, and then once monthly for 6 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group B (standard symptom management) (Active Comparator): Patients receive standard symptom management QW during standard of care radiation therapy and for 6 months after completing radiation therapy course.
  Interventions: Other: Palliative Therapy

INTERVENTIONS:
Other: Palliative Therapy — Receive standard symptom management
  Other Names: Comfort Care; PA-Palliative Therapy; palliation; Palliative; Palliative Care; Palliative Treatment; Symptom Management; Symptoms Management
  Arms: Group B (standard symptom management)
Other: Quality-of-Life Assessment — Complete quality of life questionnaire
  Other Names: Quality of Life Assessment
  Arms: Group A (quality of life questionnaire)
Other: Questionnaire Administration — Complete quality of life questionnaire
  Arms: Group A (quality of life questionnaire)

SUMMARY:
This clinical trial compares intensive symptom evaluation with supportive care to standard symptom management in patients with head and neck cancer that has not spread to other places in the body (non-metastatic). Standard symptom management involves symptom management during and after radiation therapy, using problem-focused history and physical examination followed by appropriate symptomatic management as appropriate per treating physician's discretion. Intensive symptom management with monitoring patient reported outcomes is performed among patients with metastatic cancers receiving systemic therapies and with various cancers receiving radiation therapy. This trial may help researchers determine the impact of intensive symptom surveillance in patients with non-metastatic head and neck cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Using study questionnaires to determine the impact of intensive symptom evaluation with supportive care as needed per treating physician's discretion versus standard symptom management on time to first acute care visits at 3 months.

SECONDARY OBJECTIVES:

I. Using study questionnaires to determine the impact of intensive symptom evaluation with supportive care as needed per treating physician's discretion versus standard symptom management on (1) changes in health-related quality of life (HRQOL), financial burden, and caregiver burden from baseline, (2) time to first acute care visits at 1 or 6 month, (3) locoregional (LRF) and distant failure (DF), and (4) progression-free (PFS) and overall survival (OS) outcomes.

II. Using study questionnaires to determine the impact of intensive symptom evaluation with supportive care as needed per treating physician's discretion versus standard symptom management when stratified.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP A: Patients complete a quality of life questionnaires over 10-15 minutes twice weekly (BIW) during standard of care radiation therapy and once weekly (QW) for the first month after completing standard of care radiation therapy course, and then once monthly for 6 months.

GROUP B: Patients receive standard symptom management QW during standard of care radiation therapy for 6 months after completing radiation therapy course.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Age >= 18 years of age
* PATIENTS: Diagnosed with biopsy-proven, non-metastatic squamous cell carcinoma of head and neck
* PATIENTS: Scheduled to start curative-intent radiation therapy within 4 weeks
* PATIENTS: Able to provide informed consent in English
* PATIENTS: Able to read and write in English
* PATIENTS: Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related assessment
* PATIENTS' INFORMED CAREGIVER (e.g. family members, friends): They are verbally identified by eligible patients as a caregiver
* PATIENTS' INFORMED CAREGIVER (e.g. family members, friends): They are not receiving any payment to provide care for patients
* PATIENTS' INFORMED CAREGIVER (e.g. family members, friends): Able to provide informed consent in English
* PATIENTS' INFORMED CAREGIVER (e.g. family members, friends): Able to read and write in English

Exclusion Criteria:

* PATIENTS: Diagnosed with metastatic head and neck cancer
* PATIENTS: Eligible for palliative-intent radiation therapy only
* PATIENTS: Pregnant female participants
* PATIENTS: Unwilling or unable to follow protocol requirements
* PATIENTS: Any condition which in the Investigator's opinion deems the participant an unsuitable candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Time to first acute care visit | At 3 months
  to evaluate the impact of intensive symptom evaluation compared to standard symptom management on time to first acute care visits at 3 months with time to first acute care visits.

SECONDARY OUTCOMES:
Change in Health-related quality of life EORTC QLQ-C30 | Baseline to 6 months
  Patient reported outcome assessment measured data Quality of life data will be obtained via European Organisation for Research and Treatment of Cancer Quality of Life Cancer Patients (EORTC QLQ-C30). It It is a 30-item questionnaire assessing other cancer-related symptoms
Change in financial burden | Baseline to 6 months
  Change in patient reported outcomes measured using the Comprehensive Score for Financial Toxicity (COST). Financial toxicity is assessed using an 11-item patient-reported measure of financial stress used in cancer patients. The COST yields a total score with higher scores indicating less financial toxicity
Change in caregiver burden | Baseline to 6 months
  Will be evaluated with the Caregiver Reaction Assessment (CRA). Summary score range between 5 and 120. A higher score indicates a higher level of burden.
Time to first acute care visits | At 1 or 6 month
  Patient reported 9 item questionnaire to evaluate the impact of intensive symptom evaluation compared to standard symptom management on time to first acute care visits at 3 months with time to first acute care visits.
Locoregional failure | Time interval from diagnosis to locoregional failure, assessed up to 6 months
  Analyzed with the questionnaire and standard of care tumor assessment, disease progression, and survival status information.
Distant failure | Time interval from diagnosis to distant failure outside head and neck region, assessed up to 6 months
  Analyzed with the questionnaire and standard of care tumor assessment, disease progression, and survival status information.
Progression free survival | Time interval from diagnosis to tumor recurrence or progression of disease, assessed up to 6 months
  Analyzed with the questionnaire and standard of care tumor assessment, disease progression, and survival status information.
Overall survival | Time interval from diagnosis to death from any cause, assessed up to 6 months
  Analyzed with the questionnaire and standard of care tumor assessment, disease progression, and survival status information.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag K Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States